CLINICAL TRIAL: NCT05086419
Title: Sub-symptom Threshold Aerobic Exercise Training for Patients With Exercise Intolerance and Persistent Symptoms After Mild Traumatic Brain Injury - A Randomized Controlled Trial
Brief Title: Sub-symptom Threshold Aerobic Exercise After Mild Traumatic Brain Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ingerid Kleffelgård, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK #256109
Record Dates: First submitted 2021-10-05; First posted 2021-10-20 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; Buffalo Concussion Treadmill Test; Sub-symptom aerobic exercise
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind parallel group design.
Who Masked: Outcomes Assessor
Masking Description: After written informed consent, patients will be randomized to the intervention or control group using computer-generated lists. Block randomization with variable block size that is unknown to the research group will be used. Follow-up tests at T1 and T2 will be performed by a research assistant who is blind to the group distribution and who is not involved in any parts of the intervention. Statisticians will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The exercise group will in addition to treatment as usual, receive sub-symptom threshold aerobic exercise for approx. 30 minutes 3-5x / week for 12 weeks. Sub-symptom threshold aerobic exercise is based on the individual patient's symptom threshold and will be between 80-90% of the maximum heart rate achieved during testing/BCTT. To ensure proper exercise dosage and progression, participants will be retested every 3 weeks. An experienced doctor and / or physiotherapist will carry out the testing and guide the participants in the content and dosage (duration, intensity, and frequency) of the sub-symptom threshold aerobic exercise/intervention.
  Interventions: Other: Sub-symptom threshold aerobic exercise
- Treatment as usual group (No Intervention): The treatment as usual group will receive assessment and treatment provided by a multidisciplinary outpatient rehabilitation team. Patients will undergo a medical examination and assessment of physical, cognitive and mental health and functioning, followed by individually adapted rehabilitation. The interdisciplinary team consists of a specialist in physical medicine and rehabilitation, neuropsychologist, occupational therapist, physiotherapist, and social worker. The main focus is on stabilizing the level of function in everyday life and gradual return to work and education.
  Participants receive general advice on physical activity based on recommendations from the Norwegian Directorate of Health, but not specific guidance in sub-symptom threshold aerobic exercise and help with exercise dosage (frequency, duration and intensity).

INTERVENTIONS:
Other: Sub-symptom threshold aerobic exercise — For the first three weeks, participants will be offered guided sub-symptom threshold aerobic exercise on a treadmill or exercise bike once a week. The remaining 2-4 sub-symptom threshold aerobic exercise workouts per. week will be on their own. Location and mode of exercise (treadmill, walking, jogging, exercise bike / bicycle, swimming, or elliptical machine) will be individually adapted to the patients experience, preferences and opportunities. The intensity of the sub-symptom threshold aerobic exercise will always be monitored using a heart rate monitor and/or ratings of perceived exertion (Borg RPE). If there still is a need for closer follow-up after the first three weeks, a physiotherapist in primary health care service will be involved under supervision from a physiotherapist (research fellow) in the project.
  Arms: Exercise group

SUMMARY:
This Randomized Controlled Trial (RCT) will explore the effect of sub-symptom threshold aerobic exercise on persistent post-concussion symptoms and exercise intolerance in patients with mild Traumatic Brain Injury (TBI). The hypothesis is that sub-symptom training will reduce the symptom pressure, normalize exercise tolerance, reduce patient-specific activity limitations and improve health-related quality of life. To improve the chances of conducting a high-quality RCT, a feasibility trial will be completed prior to the definitive RCT.

DETAILED DESCRIPTION:
Background: Persistent post-commotio symptoms (PCS) affect between 34% and 46% of individuals after a mild traumatic brain injury (TBI). Many also experience exercise intolerance. Sub-symptom threshold aerobic exercise (exercise at an intensity level that does not increase symptoms) is proposed as treatment both to increase the exercise tolerance and to ease the symptom burden after the injury.

Main purpose: The main purpose of this study is to evaluate whether a progressive sub-symptom threshold exercise program in addition to ordinary rehabilitation will lead to clinically meaningful improvement of symptom burden, normalize exercise tolerance, increase physical activity, improve health-related quality of life, and reduce patient-specific activity limitations compared to a control group that only receives ordinary rehabilitation.

Design: Randomized, controlled, single-blind parallel-group study with three measurement times; T0 at baseline, T1 after the intervention and T2 six months after T1.

Method: 68 patients between the ages of 18 and 60 with exercise intolerance and persistent PCS will be recruited to the study and randomized to two groups. All participants will receive ordinary rehabilitation. The intervention group will in addition receive sub-symptom threshold aerobic exercise for 12 weeks with weekly follow-up by a physiotherapist and a retest every 3 weeks for optimal dosage and progression. Rivermead post-concussion symptoms questionnaire (RPQ) will be the main outcome measure. The secondary outcome measure will be a test of exercise tolerance - the Buffalo Concussion Treadmill Test (BCTT). Other outcome measures include the patient-specific functional scale that measures patient-specific activity limitations, as well as outcome measures for health-related quality of life, anxiety and depression, specific symptoms such as dizziness, headache and fatigue, and level of physical activity.

Clinical relevance: Since people with persistent symptoms after mild TBI often have reduced level of functioning and difficulty working / studying full time, there is a great need for an individually tailored intervention that has the potential to reduce persistent symptoms and improve functioning This project will increase the evidence based knowledge about the effect of sub-symptom threshold aerobic exercise in patient with persistent symptoms after mild TBI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild TBI defined by the World Health Organization (WHO) Collaborating Center Task Force definition: 1) one or more of the following: confusion or disorientation, loss of consciousness (LOC) ≤30 minutes, post-traumatic memory loss (PTA) ≤24 hours and / or transient neurological focal deficits and intracranial lesions that do not require surgery; 2) Glasgow Coma Scale (GCS) score of 13-15 at least 30 minutes after trauma).
* 18-60 years with persistent post-commotio symptoms (minimum 3 months maximum 2 years).
* Reduced tolerance to physical activity/exercise intolerance (self-reported worsening of symptoms such as dizziness and headache during physical activity and exercise).

Exclusion Criteria:

* Other neurological or psychiatric conditions (not including anxiety and depression) listed in the medical record. Heart-lung disease, extremity injuries that prevent physical exercise, drug addiction and insufficient understanding of the Norwegian language (unable to follow instructions and/or fill in forms). Normal BCTT.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change on the Rivermead Post Concussion Symptoms Questionnaire - RPQ | 12 weeks and 6 months.
  A 16-item standardized and validated questionnaire designed to measure the severity of post-concussion symptoms following TBI. The five-point ordinal scale ranges from 0 (no problem) to 4 (severe problem). The total score ranges from 0-64, with higher scores indicating a higher symptom load. RPQ has satisfactory psychometric properties and is a widely used in TBI and persistent post-commotio symptoms research. The minimum clinically important difference (MCID) is 4.6 points.

SECONDARY OUTCOMES:
Change on the Buffalo Concussion Treadmill Test - BCTT | 12 weeks and 6 months.
  Buffalo Concussion Treadmill Test (BCTT) is a standardized test of exercise tolerance developed for patients with mild TBI/concussion. Exercise tolerance is tested by gradually increasing the load while walking on a treadmill. The test protocol starts with a speed set at 6.8 km/h at 0% incline for the first minute. The speed will be maintained but the incline will be increased by 1% every minute thereafter. Every minute, symptoms (NRS scale), ratings of perceived exertion (Borg RPE), HR and blood pressure are registered. The test is stopped by symptom exacerbation defined as an increase of ≥ 3 points on a 0-10 (best-worst) point NRS scale or at the point of voluntary exhaustion (Borg RPE scale ≥17). If the maximum incline of 15% is reached, the speed will be in increased by 0,5 km/h each subsequent minute until the stop criteria described over is reached. The test will not be performed if the patients report symptoms ≥ 7 on the NRS scale.

OTHER OUTCOMES:
Change on the Patient-specific functional scale (PSFS) | 12 weeks and 6 months.
  The Patient-specific functional scale (PSFS) is a patient-specific measure whereby the patients identify activities they are unable to perform or have difficulty in performing related to their health condition. The patients were asked to rate the current level of difficulty associated with each activity by using a Numeric Rating Scale (NRS) ranging from 0 (unable to perform the activity) to 10 (able to perform the activity with no difficulty or as before the injury).
Change on the Quality of life after brain injury - Overall Scale (QOLIBRI - OS) | 12 weeks and 6 months.
  Quality of life after brain injury (QOLIBRI) will be used to examine health-related quality of life (HRQL). The questionnaire consists of 37 questions divided into 6 dimensions of HRQL: Cognition, Self, Daily life and Autonomy, Social relationships, Emotions and Physical problems. Each item is scored on a 5-point scale, from 1 (not-at-all satisfied) to 5 (very satisfied). The total score range of 0 (lowest) to 100 (highest). A score below 60 points has been suggested as poor HRQL. The QOLIBRI is applicable to people with TBI of all severities and at all time points after the injury.
Change on the Patient Health Questionnaire (PHQ-9) | 12 weeks and 6 months.
  Patient Health Questionnaire (PHQ-9) will be used to examine/assess depressive symptoms. The questionnaire consists of 9 items on a 4 point scale ranging from 0-27 (best-worst). PHQ-9 is validated and often used in people with TBI.
Change on the Generalized Anxiety Disorder Scale (GAD-7) | 12 weeks and 6 months.
  The Generalized Anxiety Disorder Scale (GAD-7) will be used to examine anxiety. The questionnaire consists of 7 items ranging from 0-21 (best-worst).
Change on the Fatigue Severity Scale (FSS). | 12 weeks and 6 months.
  The Fatigue Severity Scale (FSS) consists of 9 questions about the physical and cognitive effects of fatigue. It is scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. The total score ranges from 9 to 63, the higher the score, the more severe fatigue.
Change on the International Physical Activity Questionnaire (IPAQ) | 12 weeks and 6 months.
  The International Physical Activity Questionnaire (IPAQ) is a 7 item questionnaire that will be used to register health-related physical activity. The response can be categorized into three categories: 1 = inactive, 2 = minimally active, 3 = Health Enhancing Physical Activity (HEPA) active.
The Problematic Experience of Therapy scale (PETS) | 12 weeks and T2 six months.
  Adherence to training will be measured with the PETS which is a brief quantitative measure developed to reflect the most commonly reported reasons for discontinuing therapy/training given by patients undergoing self-managed home-based rehabilitation/training.

CONTACTS AND LOCATIONS:
Overall Officials: Ingerid Kleffelgård, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valaas LV, Soberg HL, Rasmussen MS, Steenstrup SE, Andelic N, Kleffelgard I. Sub-symptom threshold aerobic exercise for patients with persisting post-concussion symptoms and exercise intolerance after mild traumatic brain injury - a study protocol with a nested feasibility study for a randomized controlled trial. BMC Neurol. 2023 May 3;23(1):179. doi: 10.1186/s12883-023-03221-7. PMID 37138202